CLINICAL TRIAL: NCT04416646
Title: Cabozantinib in the Elderly With Metastatic Renal Cell Carcinoma: Observational Study
Brief Title: Cabozantinib in the Elderly With Metastatic Renal Cell Carcinoma
Acronym: ZEBRA
Status: Active, not recruiting | Type: Observational
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Principal Investigator, Umberto basso, Doctor of Medicine I level, Istituto Oncologico Veneto IRCCS
Other Study IDs: ZEBRA
Record Dates: First submitted 2020-05-12; First posted 2020-06-04 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Renal Cell Carcinoma
Keywords: Cabozantinib
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cabozantinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Cabozantinib — The regimen will be a single oral dose administered daily on a continuous schedule, taken with or without food. The standard dose is 60 mg per day, which can be reduced to 40 or 20 mg according to the latest version of the Summary of Product Characteristics-SPC available. The treating oncologist will evaluate the opportunity to prudentially start treatment at 40 mg/daily in patients screening positively at G8 screening tool, and then escalate to 60 mg/daily only in case of absence of toxicity ³grade 2 at subsequent cycles. Temporary suspensions of treatment are allowed according to the local practice and will be registered if ³ 7 days.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Cabozantinib in the treatment of patients with renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 years
* Histological diagnosis of Renal Cell Carcinoma (any histology, with the exclusion of urothelial carcinomas)
* Locally advanced disease or metastatic disease (any site, measurable or non- measurable lesions), progressing after at least one line of VEGFR-targeted therapy (as per official registration of the drug at AIFA, in case of extension to first-line treatment, TKI-naïve patients will also be eligible), with or without previous exposure to check-point inhibitors.
* Life expectancy of at least 3 months
* Adequate hepatic, renal and bone marrow function as judged by the treating oncologist.
* Written informed consent

Exclusion Criteria:

* Inability to swallow cabozantinib tablets
* Serious comorbidities or cognitive impairment, which may interfere with cabozantinib administration and/or patient's follow up, as judged by the treating physician
* Absence of a reliable caregiver, as judged by the treating physician

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients will be enrolled from Italian oncology Centers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Clinical tolerability of Cabozantinib | Average of 1 year
  the main purpose is to register the Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]

SECONDARY OUTCOMES:
Description of response rate of patients treated with Cabozantinib. | From date of randomization until the date of last documented, assessed up to 18 months"
  according to RECIST criteria, only patients with measurable disease will be evaluated for response

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Oncologico Veneto, Padua, Italy

IPD SHARING:
Plan to Share IPD: Undecided